CLINICAL TRIAL: NCT00158912
Title: Ventricular Arrhythmia Suppression Trial
Brief Title: VAST - Ventricular Arrhythmia Suppression Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-CA-060903-T
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2006-11

CONDITIONS: Tachycardia
MeSH Terms: conditions — Tachycardia | interventions — Defibrillators, Implantable

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator

SUMMARY:
The purpose of VAST is to determine whether the Rate Smoothing feature in Guidant's PRIZM/VITALITY-family ICDs has an effect on the incidence of ventricular tachyarrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive a commercially available Guidant PRIZM, PRIZM 2, or VITALITY AVT ICD
* Patients who sign and date a Patient Informed Consent prior to study enrollment
* Patients who remain in the clinical care of physicians of their implanting center

Exclusion Criteria:

* Patients who have chronic atrial fibrillation. Paroxysms of AF are not an exclusion criterion, but the patient must be in normal sinus rhythm at the time of randomization. If history of AF is unknown or uncertain, or the patient was recently cardioverted, there must be at least 23 hours of normal sinus rhythm within the 24 hour period preceding randomization
* Patients who previously had an ICD
* Patients with current indications for cardiac resynchronization therapy with defibrillation (CRT-D)
* Patients whose life expectancy is less than 12 months due to other medical conditions
* Patients who are expected to receive a heart transplant during the duration of the study
* Patients who have or who are likely to receive a tricuspid or other valve prosthesis
* Patients who are currently enrolled in another investigational study of active medical therapy. Each instance should be brought to Guidant's Clinical Application Research Studies (CARS) group to determine eligibility
* Patients who are younger than 18 years of age
* Patients who are mentally incompetent and cannot give a Patient Informed Consent or participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 550
Dates: Start 2003-08; Study Completion 2005-05

PRIMARY OUTCOMES:
The primary endpoint for this study will be the number of episodes of ventricular tachyarrhythmia in each patient during each follow-up period (ON vs. OFF treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Friedman, MD, Principal Investigator — Mayo Clinic